CLINICAL TRIAL: NCT06692764
Title: A Phase II Study to Assess the Effect of AZD0780 on Ambulatory Blood Pressure in Participants With Atherosclerotic Cardiovascular Disease or Risk Equivalents and Elevated Low-Density Lipoprotein Cholesterol
Brief Title: A Study to Assess the Effect of AZD0780 on Ambulatory Blood Pressure
Acronym: AZD0780-ABPM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D7960C00009
Record Dates: First submitted 2024-10-28; First posted 2024-11-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Ambulatory Blood Pressure.; Atherosclerotic Cardiovascular Disease.; Elevated Low-density Lipoprotein Cholesterol
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Potential participants will be screened to assess their eligibility to enter the study up to 7 days prior to first administration of study intervention. Eligible participants will be randomized to Treatment Sequence AB or BA on Period 1 Day 1. A 14-day washout period will be required between the final dose in Period 1 and start of baseline ABPM in Period 2.
  In Periods 1 and 2, participants will return to the study site for an OPV on Day -1 for the start of the baseline ABPM. The ABPM device will be worn for 25 hours. Participants will return to the study site for an OPV on the following day (Day 1) for removal of the ABPM device and to begin self-administration of AZD0780 or placebo for 29 ± 2 days as per the randomization scheme. First dose of study intervention will be taken after the ABPM device is removed on Day 1 at the study site after the baseline ABPM is qualified (i.e., determined not to require repeat).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD0780 (Experimental): Following randomization to treatment sequence, participants receive AZD0780 during period 1 or 2.
  Interventions: Drug: AZD0780
- Placebo (Placebo Comparator): Following randomization to treatment sequence, participants receive Placebo during period 1 or 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 0 mg (Placebo). Participants will receive three bottles, each containing 35 tablets with placebo tablets.
  Participants will take 1 tablet from each bottle on each scheduled day of study intervention, which will provide the placebo dose.
  Arms: Placebo
Drug: AZD0780 — Dose 1 Participants will receive three bottles, each containing 35 tablets:
  * 1 bottle of dose a AZD0780 tablets
  * 1 bottle of dose b AZD0780 tablets
  * 1 bottle of dose c AZD0780 tablets Participants will take 1 tablet from each bottle on each scheduled day of study intervention, which will provide the AZD0780 dose.
  Arms: AZD0780

SUMMARY:
This is a Phase II, multi-centre, randomized, double-blind, placebo-controlled, crossover study to evaluate the effect of AZD0780 Dose 1 versus placebo on systolic blood pressure (SBP) at Week 4, as measured by 24-hour ambulatory blood pressure monitoring (ABPM) in participants with ASCVD or risk equivalents and LDL-C ≥ 70 mg/dL, on stable medication.

DETAILED DESCRIPTION:
This is a Phase II, multi-centre, randomized, double-blind, placebo-controlled, crossover study to evaluate the effect of AZD0780 Dose 1 versus placebo on systolic blood pressure (SBP) at Week 4, as measured by 24-hour ambulatory blood pressure monitoring (ABPM) in participants with ASCVD or risk equivalents and LDL-C ≥ 70 mg/dL, on stable medication.

Approximately 30 sites in the United Sites will enroll adult participants with Atherosclerotic Cardiovascular Disease or Risk Equivalents and Elevated Low-density Lipoprotein Cholesterol.

Eligible participants will be randomized (1:1) on Period One (1) Day One (1) to One (1) of Two (2) treatment sequences.

Potential participants will be screened to assess their eligibility to enter the study up to 7 days prior to first administration of study intervention. Eligible participants will be randomized to Treatment Sequence AB or BA on Period One (1) Day One (1). A 14-day washout period will be required between the final dose in Period One (1) and start of baseline ABPM in Period Two (2).

In Periods One (1) and Two (2), participants will return to the study site for an outpatient visit (OPV) on Day -1 for the start of the baseline ABPM. The ABPM device will be worn for 25 hours. Participants will return to the study site for an OPV on the following day (Day 1) for removal of the ABPM device and to begin self-administration of AZD0780 or placebo for 29 ± 2 days as per the randomization scheme. First dose of study intervention will be taken after the ABPM device is removed on Day 1 at the study site after the baseline ABPM is qualified (i.e., determined not to require repeat). Additional OPVs will be required on Days 14 (± 2 days), 28 (± 2 days), and 29 (day after Day 28 [± 2 days]). On Days 28 and 29 of each period, the ABPM device will be worn for 25 hours. Study intervention will continue to be taken on each day after the start of Week 4 (Days 28 and 29) 24-hour ABPM for Periods 1 and 2 until a qualified ABPM is obtained. Only 1 repeat may be attempted within 2 days of the end of the first ABPM attempt. Participants will return to the study site for a follow-up visit 14 (± 2) days after the last dose of study intervention in Period Two (2).

Serial pharmacokinetic blood samples will be collected predose and up to 7 hours postdose on Day 14 and predose on Day 28 in each period. Monitoring of adverse events, vital sign measurements, 12-lead electrocardiograms, clinical laboratory tests, and physical examinations will be performed to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age at the time of signing the informed consent.
2. Participants with a history of ASCVD defined as myocardial infarction, stroke, or symptomatic peripheral arterial disease, or with risk factors hereof.
3. Participants with a fasting serum LDL-C ≥ 70 mg/dL (1.8 mmol/L) at screening.
4. Should be receiving stable SoC therapy for their comorbidities for at least 4 weeks prior to screening. There should be no planned medication or dose changes during study participation.
5. Body mass index ≥ 19.0 kg/m2.
6. Sex: males and females (females of non-childbearing potential).

Exclusion Criteria

1. eGFR < 45 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration creatinine equation (2021) at screening.
2. History or presence of gastrointestinal, hepatic, or renal disease, or any other conditions known to interfere with absorption, distribution, metabolism, or excretion of drugs.

4. Poorly controlled type 2 diabetes mellitus, defined as HbA1c > 10% at screening.

5. Participants with history of coronary artery bypass graft surgery ≤ 6 months prior to screening or percutaneous coronary intervention ≤ 3 months prior to screening.

6. Heart failure with New York Heart Association Class III to IV. 9. Low-density protein or plasma apheresis within 12 months prior to Period 1 Day -1.

10. Uncontrolled hypertension defined as average of triplicate seated SBP > 160 mmHg or DBP > 90 mmHg at screening.

11. Pulse rate after 10 minutes seated rest < 50 or > 100 bpm at screening. 12. Any laboratory values with the following deviations at screening; test may be repeated at the discretion of the investigator if abnormal:

(a) Any positive result on screening for hepatitis B, hepatitis C, or HIV; (b) ALT > 1.5 × ULN; (c) AST > 1.5 × ULN; (d) TBL > ULN; (e) Haemoglobin < 12 g/dL in males or < 11 g/dL in females; (f) Potassium < lower limit of normal. 13. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as judged by the investigator, including:

1. family history of long QT syndrome;
2. PR interval prolongation > 240 ms;
3. QTcF > 450 ms; (> 470 ms in participants with bundle branch block)
4. any intermittent or persistent high degree atrioventricular-block grade II-III and sinus node dysfunction with significant sinus pause untreated with pacemaker; and cardiac tachyarrhythmias requiring treatment.

   18. Lomitapide within 12 months prior to Period 1 Day -1. 19. Current or previous treatment with drugs for reduction or inhibition of PCSK9 (approved or investigational, eg, evolocumab, alirocumab, or inclisiran) within 12 months prior to Period 1 Day -1.

   20. Fibrate therapy and derivatives are prohibited. 21. Receiving or has received within 14 days of screening, medication that contains a black box warning for significant QT prolongation. A list of prohibited medications can be found in Appendix G.

   22. Nutraceuticals or homeopathic treatments which may have an impact on BP. 26. Participants working 3rd shift or night shifts based on potential changes in circadian rhythm.

   27. Participants with sleep disorders that would affect ABPM measurements, in the investigator's opinion.

   28. Participant arm circumference not appropriate for available ABPM cuff circumference, or participant has a medical device (eg, continuous glucose monitor) that prevents use of the ABPM device, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory 24-hour average SBP at Week 4 | Week 4
  Change from baseline in ambulatory 24-hour average systolic blood pressure (SBP) at Week 4

SECONDARY OUTCOMES:
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory 24-hour average DBP at Week 4 | Week 4
  Change from baseline in ambulatory 24-hour average diastolic blood pressure (DBP) at Week 4
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory nighttime average SBP at Week 4 | 4 Weeks
  Change from baseline in ambulatory nighttime average systolic blood pressure (SBP) at Week 4
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory daytime average SBP at Week 4 | 4 Weeks
  Change from baseline in ambulatory daytime average systolic blood pressure (SBP) at Week 4
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory nighttime average DBP at Week 4 | 4 Weeks
  Change from baseline in ambulatory nighttime average diastolic blood pressure (DBP) at Week 4
To assess the effect of treatment with AZD0780 dose 1 versus placebo on ambulatory daytime average DBP at Week 4 | 4 Weeks
  Change from baseline in ambulatory daytime average diastolic blood pressure (DBP) at Week 4

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Research Site, Inglewood, California
  - Research Site, Northridge, California
  - Research Site, Pomona, California
  - Research Site, Boca Raton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Potomac, Maryland
  - Research Site, New Bedford, Massachusetts
  - Research Site, New Windsor, New York
  - Research Site, Beavercreek, Ohio
  - Research Site, Horsham, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Hurst, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Paris, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/